CLINICAL TRIAL: NCT03010618
Title: Hall Teknik Ile Uygulanan Paslanmaz Celik kronların Okluzal Dikey Boyuta Etkilerinin değerlendirilmesi
Brief Title: The Effects of Stainless Steel Crowns Applied With Hall Technique on Occlusal Vertical Dimension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Sarp Kaya, Specialist, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6.2016/45
Record Dates: First submitted 2016-12-31; First posted 2017-01-05 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Caries, Dental
Keywords: hall technique; stainless steel crowns; temporomandibular joint; dental caries; occlusion
MeSH Terms: conditions — Dental Caries; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Other)
  Interventions: Other: Hall technique stainless steel crowns

INTERVENTIONS:
Other: Hall technique stainless steel crowns — Primary carious tooth will be treated with stainless steel crowns without local anesthesia or caries removal and the increase in the occlusal vertical dimension will be monitored in two subsequent appointments with measuring canine overbite.

SUMMARY:
In recent years restoring carious of fractured primary teeth with stainless steel crowns (SSC) has became more popular than ever. On the other hand the traditional operative approach of complete removal of caries is steadily losing support due to successful results with materials of high microleakage resistance.

Treatment time and pain control in asymptomatic teeth has always been a problem in children. Hall technique is a minimally invasive treatment protocol that doesn't require local anesthesia, use of rotating devices for caries removal to restore primary teeth with SSC.

But this protocol also raised questions in the scientific community about its possible effects on the dentition and temporomandibular joint (TMJ) for causing primary occlusal contact and increasing vertical dimension.

The aim of our research is to study the effects of Hall technique's premature occlusal contact on TMJ.

ELIGIBILITY:
Inclusion Criteria:

* No systemical illness
* Willing to come to control appointments
* No symptoms of pulpal inflammation
* To have at least 1, 3 at most dentin caries primary teeth without infection, mobility, Angle class I profile and molar relation
* Willing to participate the study

Exclusion Criteria:

* History of diagnosed systemic illness
* Anterior/ posterior crossbite
* Presence of dental pain
* Root resorption exceeding 2/3's of the treated tooth
* Gingival inflammation, periodontal disease
* Signs of parafunctionism, bruxism
* Facial asymmetry
* Signs or symptoms of temporomandibular disfunction
* Not willing to participate

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete canine overbite return | 30 days
  The length of overbite between upper and lower canines will be measured at beginning of the study with marking the overlapping contact point of the upper left canine and length of a straight line to the tip of the lower left canine will be recorded in mm with a standard WHO gingival probe. Full return to this level will be considered as "Complete canine overbite return" and failure to reach this level will in 30 days will require the patient to be scheduled for an extra recall in every 2 weeks until overbite returns to the pretreatment level.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Faculty of Dentistry Department of Pediatric Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] Innes NP, Stirrups DR, Evans DJ, Hall N, Leggate M. A novel technique using preformed metal crowns for managing carious primary molars in general practice - a retrospective analysis. Br Dent J. 2006 Apr 22;200(8):451-4; discussion 444. doi: 10.1038/sj.bdj.4813466. PMID 16703041
- [Background] Kindelan SA, Day P, Nichol R, Willmott N, Fayle SA; British Society of Paediatric Dentistry. UK National Clinical Guidelines in Paediatric Dentistry: stainless steel preformed crowns for primary molars. Int J Paediatr Dent. 2008 Nov;18 Suppl 1:20-8. doi: 10.1111/j.1365-263X.2008.00935.x. PMID 18808544
- [Result] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Result] Gallagher S, O'Connell BC, O'Connell AC. Assessment of occlusion after placement of stainless steel crowns in children - a pilot study. J Oral Rehabil. 2014 Oct;41(10):730-6. doi: 10.1111/joor.12196. Epub 2014 Jun 10. PMID 24913609